CLINICAL TRIAL: NCT04287205
Title: The Effect of Dydrogesterone on Sexual Function in Women With Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: endo-fsfi
Record Dates: First submitted 2020-02-23; First posted 2020-02-27 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Endometriosis; Sexual Dysfunction
MeSH Terms: conditions — Endometriosis; Sexual Dysfunction, Physiological | interventions — Dydrogesterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- women with endometriosis (Experimental)
  Interventions: Drug: Dydrogesterone

INTERVENTIONS:
Drug: Dydrogesterone — 79 women, aged between 18 and 45 years, who were examined at our tertiary gynecology outpatient clinic between April 2019 and March 2020, with surgically diagnosed endometriosis, were included in this study. They received a treatment with 5 mg dydrogesterone administered orally twice daily for 21 days; from the 5th to 25th day of each menstrual cycle, for a total of 6 months. They were evaluated pre- and posttreatment in terms of their age, parity, and body mass index (BMI). Female Function Sexual Index (FSFI) and visual analogue scale (VAS) scores were recorded pre- and posttreatment

SUMMARY:
This study aimed to assess the effects of dydrogesterone on sexual function in women with endometriosis using Female Function Sexual Index (FSFI).

DETAILED DESCRIPTION:
Sexual dysfunction is an important outcome for patients with endometriosis. In this study, we compare the fsfi (female sexual function index) questions and the scores before and after dydrogesterone treatment in patients with endometriosis. We aim to measure the effect of dydrogesterone in patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* no history of malignancies,
* normal findings at gynecological examinations and transvaginal ultrasonography
* normal uterine size, normal cervical smear results,
* patients not use any contraception methods in the last 6 months

Exclusion Criteria:

* with a history of systemic and/or psychiatric diseases,
* gynecological pathologies (myoma uteri, endometriosis, uterine anomalies, existing genital infections)
* pelvic organ prolapse
* pelvic surgeries

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 79 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
The Effect of Dydrogesterone on Sexual Function | 6 months
  In this study, we compare the fsfi(female sexual function index) questions and the scores before and after dihydrogestreone treatment in patients with endometriosis. We aim to measure the effect of dihydrogesterone in patients with endometriosis.

SECONDARY OUTCOMES:
The Effect of Dydrogesterone on Sexual Function in women with endometrioma | 6 months
  In this study, we compare the fsfi(female sexual function index) questions and the scores before and after dihydrogestreone treatment in patients with endometriosis. We aim to measure the effect of dihydrogesterone in patients with endometriosis.(with and without endometrioma)

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes